CLINICAL TRIAL: NCT05400057
Title: the Oncogenic Potential of Salivary miRNA-93 and miRNA-412-3P in Oral Lichen Planus Patients
Status: Completed | Type: Observational
Sponsor: Moataz Mahmoud (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Moataz Mahmoud, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 6222
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Oral Lichen Planus; Oral Cancer
Keywords: miRNA; Oral Lichen Planus; Oral Cancer
MeSH Terms: conditions — Lichen Planus, Oral; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: Oral Lichen Planus patients. Patients will be diagnosed clinically and histologically.
- Group 2: Healthy patients. Patients without any systemic or oral lesions, not taking drugs for at least the the last 6 months
- Group 3: Oral Squamous Cell Carcinoma

SUMMARY:
Assessment The oncogenic potential of salivary microRNA-93 and microRNA-412-3p in oral lichen planus

DETAILED DESCRIPTION:
Oral lichen planus is one of the most common prevalent muco-cutaneous chronic diseases. The disease is definitely auto-immune type .Despite having idiopathic etiology, many risk factors can be considered including systemic diseases, psychogenic diseases, dental restorations and some drugs.

The oral lesions are mainly bilateral, with frequent appearance in the inner buccal mucosa. It can be categorized into three forms; reticular form, atrophic form and bullous-erosive form.

The disease is considered as premalignant lesion as it has high potential of malignant transformation. T-lymphocytes infiltration in the basal cell layer of the epithelium and cytoid bodies are characteristic histopathologic features of the disease.

MicroRNAs (miRNAs) are endogenous short non-coding about 22 nucleotides RNAs in length. They perform major regulatory roles by targeting messenger RNAs (mRNAs) for cleavage or translational repression in animals and plants. they comprise one of the classes of gene regulatory molecules and definitely impact the output of many genes coding protein.

Previous studies have reported their critical role in development of various diseases in broad pathological conditions. Numerous studies have investigated the expression of miRNAs as diagnostic and prognostic biomarkers in potentially malignant diseased patients from human specimens, confirming these miRNAs as risk biomarkers for malignant transformation with excellent results.

miRNAs might make contribution as biomarkers for risk of development, for prognosis and response to treatment of oral cancer. Some studies have examined miRNA in Oral Lichen Planus (OLP) patients, not all of the have shown significant difference in miRNA changes, the role of miRNAs in malignant transformation of OLP is under examination.

MiR-93 is type of miRNAs within the miR-106b∼25 cluster. It has been reported that miRNA reinforced cell survival, corroborated sphere formation, amplified tumour growth, raised angiogenesis by enhancing endothelial cell activities and prevented apoptosis by targeting integrin-β8, a cell death-inducing antigen. These data suggested that miR-93 had important roles in carcinogenesis. Additionally, overexpression of miR-93 has been found in a broad range of cancers, including neuro-blastoma, non-small cell lung cancer, breast cancer and ovarian cancer. Furthermore, a significant increase in expression of miR-93has been detected in the saliva of OSCC patients compared to non-diseased participants. MiR-412-3p is beneficial in predicting cancer, focusing grave implications in cancer progression, and miR-412-3p was manifested to be highly expressed in extracellular vesicles from oral squamous cell carcinoma (OSCC) patients. MiRNA-93 and miRNA412-3p haven't been yet, according to our knowledge, experimented in Oral Lichen Planus patients, and they have been already assessed in OSCC patients. So, in our study, we assess the oncogenic potential of miR-93 and miR-412-3p in oral lichen patients, for more information about potential new tumour markers in Oral Lichen Planus.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age range from 40 to 70 years.
* Clinically diagnosed and histologically confirmed as having symptomatic OLP.
* Patients who agree to sign a written consent after understanding the nature of the study

Exclusion Criteria:

* -Systemic and/or local systemic drug therapy within the last 3 months prior to the start of the study
* Patients on steroidal or non-steroidal anti-inflammatory drugs (NSAIDs) for at least the last 6 months
* Patients on Retinoid, green tea supplements or another natural products therapy
* Patients with already diagnosed malignant lesion/lesions
* Pregnant or Lactating females
* Vulnerable groups as prisoners, mentally disabled, etc…

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be chosen clinically by taking patient history and clinical examination for all patients and histologically by taking incisional biopsy from the oral lesion to confirm the diagnosis of Oral Lichen Planus.
  Controls will be chosen without any oral systemic or oral lesions for accurate assessment and comparison of microRNA-93 and microRNA-412-3p between cases and controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
miRNA-93 | 2 years
  MicroRNA 93 is a functional RNA and a microRNA that in humans is encoded by the MIR93 (MicroRNA 93) gene
miRNA-412-3P | 2 years
  microRNAs (miRNAs) are short (20-24 nt) non-coding RNAs that are involved in post-transcriptional regulation of gene expression in multicellular organisms by affecting both the stability and translation of mRNAs

CONTACTS AND LOCATIONS:
Overall Officials: Moataz Taha, PhD student, Study Director — Faculty of Dentistry, CairoU; Weam Rashwan, Professor, Principal Investigator — Faculty of Dentistry, CairoU; Olfat Shaker, Professor, Study Chair — Faculty of Medicine, CairoU; Inas Abdou, Lecturer, Study Director — Center Of Radiation Oncology & Nuclear Medicine, CairoU
Locations (1):
- Facuty of Dentistry, CairoU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided